CLINICAL TRIAL: NCT02195479
Title: A Phase 3, Randomized, Controlled, Open-label Study of VELCADE (Bortezomib) Melphalan-Prednisone (VMP) Compared to Daratumumab in Combination With VMP (D-VMP), in Subjects With Previously Untreated Multiple Myeloma Who Are Ineligible for High-dose Therapy
Brief Title: A Study of Combination of Daratumumab and Velcade (Bortezomib) Melphalan-Prednisone (DVMP) Compared to Velcade Melphalan-Prednisone (VMP) in Participants With Previously Untreated Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104761; 54767414MMY3007 (Other: Janssen Research and Development, LLC); 2014-002272-88 (EudraCT Number)
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; Velcade; Melphalan; Prednisone; Daratumumab
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm A (VMP Alone) (Active Comparator): Participants will receive velcade (bortezomib) 1.3 milligram per square meter (mg/m^2) as subcutaneous injection, twice weekly at Weeks 1, 2, 4 and 5 in Cycle 1 followed by once weekly at Weeks 1, 2, 4 and 5 in Cycles 2 to 9, melphalan 9 mg/m^2 , orally, once daily (on Days 1-4) and prednisone 60 mg/m^2, orally, once daily, on Days 1 to 4 of each cycle up to Cycle 9.
  Interventions: Drug: Velcade; Drug: Melphalan; Drug: Prednisone
- Treatment Arm B (D-VMP) (Experimental): Participants will receive velcade 1.3 mg/m^2 as SC injection, twice weekly at Weeks 1, 2, 4 and 5 in Cycle 1 followed by once weekly at Weeks 1, 2, 4 and 5 in Cycles 2 to 9, melphalan 9 mg/m^2, orally, once daily (on Days 1-4) and prednisone 60 mg/m^2, orally, once daily, on Days 1 to 4 of each cycle up to Cycle 9. In addition participants will also receive daratumumab 16 mg/kg as IV infusion, once weekly, for 6 weeks in Cycle 1 and then every 3 weeks, in Cycle 2 to 9 and thereafter, once every 4 weeks until documented progression, unacceptable toxicity, or until the end of study. On days when daratumumab is given, dexamethasone 20 mg IV or PO is given 1 hour or less prior to daratumumab administration as pre medication and prednisone substitute, and prednisone 60 mg/m2 once daily will be given on Days 2-4. Following amendment 7, participants will have the option to switch to daratumumab subcutaneous (SC) on Day 1 of any cycle, at the discretion of the investigator.
  Interventions: Drug: Velcade; Drug: Melphalan; Drug: Prednisone; Drug: Daratumumab IV; Drug: Dexamethasone; Drug: Daratumumab SC

INTERVENTIONS:
Drug: Velcade — Participants will receive velcade 1.3 mg/m^2, as subcutaneous injection, twice weekly at Weeks 1, 2, 4 and 5 in Cycle 1 followed by once weekly at Weeks 1, 2, 4 and 5 in Cycles 2 to 9.
Drug: Melphalan — Participants will receive melphalan 9 mg/m^2, orally, once daily on Days 1 to 4 of each cycle up to Cycle 9.
Drug: Prednisone — Participants will receive prednisone 60 mg/m^2, orally, once daily, on Days 1 to 4 of each cycle up to Cycle 9.
Drug: Daratumumab IV — Participants will receive daratumumab 16 mg/kg as intravenous infusion, once weekly, for 6 weeks in Cycle 1 and then once every 3 weeks, in Cycle 2 to 9 and thereafter, once every 4 weeks until documented progression, unacceptable toxicity, or until the end of study .
  Arms: Treatment Arm B (D-VMP)
Drug: Dexamethasone — Participants administered with dexamethasone 20 mg IV or PO is given 1 hour or less prior to daratumumab administration as pre medication and prednisone substitute.
  Arms: Treatment Arm B (D-VMP)
Drug: Daratumumab SC — Daratumumab SC will be administered by SC injection at a fixed dose of 1800 mg once every 4 weeks until documented progression, unacceptable toxicity, or until the end of study. Following amendment 7, participants can switch from daratumumab IV to daratumumab SC.
  Arms: Treatment Arm B (D-VMP)

SUMMARY:
The purpose of this study is to determine if the addition of daratumumab to velcade (bortezomib) melphalan-prednisone (VMP) will prolong progression-free survival (PFS) compared with VMP alone in participants with previously untreated multiple myeloma who are ineligible for high dose chemotherapy and autologous stem cell transplant (ASCT).

DETAILED DESCRIPTION:
The study consists of 3 phases: Screening Phase (within 21 days prior to randomization), Treatment Phase (Cycle 1 Day 1 to discontinuation of all study treatment), and Follow-up Phase (from discontinuation of all study treatment up to death, lost to follow up, withdrawal of consent, or the study ends, whichever occurs first). Treatment phase will include 2 treatments (Treatment A: participants will receive Velcade MelphalanPrednisone (VMP) alone and Treatment B: participants will receive daratumumab in combination with VMP).Two interim analyses are planned. The first will be to evaluate safety after a total of approximately 100 participants have been treated for at least 2 cycles or discontinued the study treatment. The second will be to evaluate cumulative interim safety and efficacy data, and will be performed when approximately 216 PFS events have been accumulated. The final OS analysis will occur when approximately 382 deaths have occurred. Efficacy will be primarily measured by comparison of PFS between the two treatment arms. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have documented multiple myeloma satisfying the calcium elevation, renal insufficiency, anemia, and bone abnormalities (CRAB) diagnostic criteria, monoclonal plasma cells in the bone marrow greater than or equal to 10 percent (%) or presence of a biopsy proven plasmacytoma, and measurable secretory disease, as assessed by the central laboratory, and defined in protocol
* Participants who are newly diagnosed and not considered candidate for high-dose chemotherapy with stem cell transplantation (SCT) due to: being age >=65 years, or in participants <65 years: presence of important comorbid conditions likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Meet the clinical laboratory criteria as specified in the protocol
* A woman of childbearing potential must have a negative serum pregnancy test at screening within 14 days prior to randomization
* Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin prior to dosing. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy

Exclusion Criteria:

* Participant has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma
* Participant has a diagnosis of Waldenstrom's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Participant has prior or current systemic therapy or SCT for multiple myeloma, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for 4 days) of corticosteroids before treatment
* Participant has peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the national cancer institute common terminology criteria for adverse events (NCI CTCAE) Version 4
* Participant has a history of malignancy (other than multiple myeloma) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years)
* Participant has had radiation therapy within 14 days of randomization
* Participant has had plasmapheresis within 28 days of randomization
* Participant has known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume in 1 second [FEV1] <50% of predicted normal), known moderate or severe persistent asthma within the last 2 years or currently has uncontrolled asthma of any classification (controlled intermittent asthma or controlled mild persistent asthma is allowed)
* Participants with known or suspected COPD must have a FEV1 test during screening
* Participant is known to be seropositive for human immunodeficiency virus (HIV), known to have hepatitis B surface antigen positivity, or history of to have a history of hepatitis C
* Participant has any concurrent medical or psychiatric condition or disease (example active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (160):
- United States (10):
  - California City, California
  - Corona, California
  - Fountain Valley, California
  - Los Angeles, California
  - Hialeah, Florida
  - Orange Park, Florida
  - Chicago, Illinois
  - Springfield, Missouri
  - Cleveland, Ohio
  - Fredericksburg, Virginia
- Argentina (4):
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Córdoba
  - Santa Fe
- Australia (9):
  - Adelaide
  - Bendigo
  - Camperdown
  - Geelong
  - Gosford
  - Greenslopes
  - Hobart
  - North Adelaide
  - Parkville
- Belgium (8):
  - Antwerp
  - Brussels
  - Charleroi
  - Ghent
  - Kortrijk
  - Roeselare
  - Turnhout
  - Yvoir
- Brazil (9):
  - Barretos
  - Cuiaba - Mount
  - Fortaleza
  - Goiânia
  - Natal
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - São Paulo
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
  - Vratsa
- Croatia (2):
  - Zadar
  - Zagreb
- Czechia (5):
  - Brno
  - Hradec Králové
  - Olomouc
  - Ostrava-Poruba
  - Prague
- Tbilisi, Georgia
- Germany (7):
  - Berlin
  - Dortmund
  - Karlsruhe
  - Potsdam
  - Saarbrücken
  - Stuttgart
  - Würzburg
- Greece (4):
  - Athens
  - Athens Attica
  - Pátrai
  - Thessaloniki
- Hungary (4):
  - Budapest
  - Debrecen
  - Kaposvár
  - Pécs
- Japan (17):
  - Chiba
  - Hitachi
  - Kanazawa
  - Kawasaki
  - Kobe
  - Kurume
  - Matsuyama
  - Nagoya
  - Narita
  - Ohgaki
  - Okayama
  - Osaka
  - Sendai
  - Shibukawa
  - Shibuya City
  - Tachikawa
  - Toyohashi
- Skopje, North Macedonia
- Poland (11):
  - Bialystok
  - Bydgoszcz
  - Chorzów
  - Gdansk
  - Legnica
  - Lublin
  - Opole
  - Słupsk
  - Warsaw
  - Warszawa Ul
  - Wroclaw
- Portugal (2):
  - Lisbon
  - Porto
- Romania (3):
  - Brasov
  - Bucharest
  - Iași
- Russia (9):
  - Arkhangelsk
  - Dzerzhinsk
  - Nizhny Novgorod
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Sochi
  - Volgograd
  - Yekaterinburg
- Serbia (5):
  - Belgrade
  - Kamenitz
  - Niš
  - Novi Sad
  - Zemun
- South Korea (6):
  - Busan
  - Gyeonggi-do
  - Hwasun
  - Incheon
  - Seongnam
  - Seoul
- Spain (16):
  - Andalucía
  - Badalona
  - Barcelona
  - Córdoba
  - Girona
  - Madrid
  - Marañón
  - Murcia
  - Ourense
  - Pamplona
  - Salamanca
  - San Cristóbal de La Laguna
  - Seville
  - Toledo
  - Valencia
  - Zaragoza
- Turkey (Türkiye) (7):
  - Altındağ
  - Ankara
  - Aydin
  - Izmir
  - Kayseri
  - Samsun
  - Tekirdağ
- Ukraine (7):
  - Cherkassy
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Khmelnitskiy
  - Lviv
  - Zaporizhzhia
- United Kingdom (8):
  - Birmingham
  - Cambridge
  - Colchester
  - Harlow
  - Leicester
  - London
  - Manchester
  - Woolwich

REFERENCES:
- [Derived] Mateos MV, San-Miguel J, Cavo M, Suzuki K, Jakubowiak A, Knop S, Doyen C, Lucio P, Nagy Z, Pour L, Grosicki S, Crepaldi A, Liberati AM, Campbell P, Yoon SS, Iosava G, Fujisaki T, Garg M, Ngo M, Katz EG, Krevvata M, Bolyard K, Carson R, Borgsten F, Dimopoulos MA. Bortezomib, melphalan, and prednisone with or without daratumumab in transplant-ineligible patients with newly diagnosed multiple myeloma (ALCYONE): final analysis of an open-label, randomised, multicentre, phase 3 trial. Lancet Oncol. 2025 May;26(5):596-608. doi: 10.1016/S1470-2045(25)00018-X. Epub 2025 Apr 9. PMID 40220771
- [Derived] Mateos MV, Dimopoulos MA, Cavo M, Suzuki K, Knop S, Doyen C, Lucio P, Nagy Z, Pour L, Grosicki S, Crepaldi A, Liberati AM, Campbell P, Yoon SS, Iosava G, Fujisaki T, Garg M, Iida S, Blade J, Ukropec J, Pei H, Van Rampelbergh R, Kudva A, Qi M, San-Miguel J. Daratumumab Plus Bortezomib, Melphalan, and Prednisone Versus Bortezomib, Melphalan, and Prednisone in Transplant-Ineligible Newly Diagnosed Multiple Myeloma: Frailty Subgroup Analysis of ALCYONE. Clin Lymphoma Myeloma Leuk. 2021 Nov;21(11):785-798. doi: 10.1016/j.clml.2021.06.005. Epub 2021 Jun 18. PMID 34344638
- [Derived] Cavo M, San-Miguel J, Usmani SZ, Weisel K, Dimopoulos MA, Avet-Loiseau H, Paiva B, Bahlis NJ, Plesner T, Hungria V, Moreau P, Mateos MV, Perrot A, Iida S, Facon T, Kumar S, van de Donk NWCJ, Sonneveld P, Spencer A, Krevvata M, Heuck C, Wang J, Ukropec J, Kobos R, Sun S, Qi M, Munshi N. Prognostic value of minimal residual disease negativity in myeloma: combined analysis of POLLUX, CASTOR, ALCYONE, and MAIA. Blood. 2022 Feb 10;139(6):835-844. doi: 10.1182/blood.2021011101. PMID 34289038
- [Derived] San-Miguel J, Avet-Loiseau H, Paiva B, Kumar S, Dimopoulos MA, Facon T, Mateos MV, Touzeau C, Jakubowiak A, Usmani SZ, Cook G, Cavo M, Quach H, Ukropec J, Ramaswami P, Pei H, Qi M, Sun S, Wang J, Krevvata M, DeAngelis N, Heuck C, Van Rampelbergh R, Kudva A, Kobos R, Qi M, Bahlis NJ. Sustained minimal residual disease negativity in newly diagnosed multiple myeloma and the impact of daratumumab in MAIA and ALCYONE. Blood. 2022 Jan 27;139(4):492-501. doi: 10.1182/blood.2020010439. PMID 34269818
- [Derived] Knop S, Mateos MV, Dimopoulos MA, Suzuki K, Jakubowiak A, Doyen C, Lucio P, Nagy Z, Usenko G, Pour L, Cook M, Grosicki S, Crepaldi A, Liberati AM, Campbell P, Shelekhova T, Yoon SS, Losava G, Fujisaki T, Garg M, Wang J, Wroblewski S, Kudva A, Gries KS, Fastenau J, San-Miguel J, Cavo M. Health-related quality of life in patients with newly diagnosed multiple myeloma ineligible for stem cell transplantation: results from the randomized phase III ALCYONE trial. BMC Cancer. 2021 Jun 2;21(1):659. doi: 10.1186/s12885-021-08325-2. PMID 34078314
- [Derived] Mateos MV, Cavo M, Blade J, Dimopoulos MA, Suzuki K, Jakubowiak A, Knop S, Doyen C, Lucio P, Nagy Z, Pour L, Cook M, Grosicki S, Crepaldi A, Liberati AM, Campbell P, Shelekhova T, Yoon SS, Iosava G, Fujisaki T, Garg M, Krevvata M, Chen Y, Wang J, Kudva A, Ukropec J, Wroblewski S, Qi M, Kobos R, San-Miguel J. Overall survival with daratumumab, bortezomib, melphalan, and prednisone in newly diagnosed multiple myeloma (ALCYONE): a randomised, open-label, phase 3 trial. Lancet. 2020 Jan 11;395(10218):132-141. doi: 10.1016/S0140-6736(19)32956-3. Epub 2019 Dec 10. PMID 31836199
- [Derived] Mateos MV, Dimopoulos MA, Cavo M, Suzuki K, Jakubowiak A, Knop S, Doyen C, Lucio P, Nagy Z, Kaplan P, Pour L, Cook M, Grosicki S, Crepaldi A, Liberati AM, Campbell P, Shelekhova T, Yoon SS, Iosava G, Fujisaki T, Garg M, Chiu C, Wang J, Carson R, Crist W, Deraedt W, Nguyen H, Qi M, San-Miguel J; ALCYONE Trial Investigators. Daratumumab plus Bortezomib, Melphalan, and Prednisone for Untreated Myeloma. N Engl J Med. 2018 Feb 8;378(6):518-528. doi: 10.1056/NEJMoa1714678. Epub 2017 Dec 12. PMID 29231133

RESULTS

PARTICIPANT FLOW:
Groups:
- Velcade, Melphalan and Prednisone (VMP): Participants received Velcade (bortezomib) 1.3 milligrams per square meter (mg/m^2) as subcutaneous (SC) injection, twice weekly at Weeks 1, 2, 4 and 5 in Cycle 1 followed by once weekly at Weeks 1, 2, 4 and 5 in Cycles 2 to 9, melphalan 9 mg/m^2 orally once daily on Days 1 to 4 and prednisone 60 mg/m^2 orally once daily on Days 1 to 4 of each cycle up to Cycle 9. Each treatment cycle was of 6 weeks. After completion of treatment, participants entered follow-up phase and were not started on subsequent anti-myeloma therapy without confirmed disease progression (assessed by the International Myeloma Working Group [IMWG] criteria). After implementation of Amendment 7, post interim overall survival (OS) analysis, sponsor confirmation of disease progression was no longer required prior to initiation of subsequent anti-myeloma therapy, except for participants who progressed on VMP arm and requested subsequent therapy with daratumumab.
- Daratumumab, Velcade, Melphalan and Prednisone (D-VMP): Participants received Velcade 1.3 mg/m^2 as SC injection, twice weekly at Weeks 1, 2, 4 and 5 in Cycle 1 followed by once weekly at weeks 1, 2, 4 and 5 in Cycles 2 to 9, melphalan 9 mg/m^2, orally once daily on Days 1 to 4 and prednisone 60 mg/m^2, orally once daily on Days 2 to 4 of each cycle up to Cycle 9. In addition, participants also received daratumumab 16 milligrams per kilogram (mg/kg) as intravenous (IV) infusion once weekly for 6 weeks in Cycle 1 and then once every 3 weeks in Cycle 2 to 9 and thereafter, once every 4 weeks (post-VMP treatment phase) until documented progression, unacceptable toxicity, or study end. On Day 1 of each cycle, dexamethasone 20 mg IV or per oral (PO) was given 1 hour or less prior to daratumumab infusion as pre-medication and prednisone substitute. Each treatment cycle was of 6 weeks. After implementation of Amendment 7, participants who were ongoing with daratumumab IV treatment were given an option to switch to daratumumab SC injection on Day 1 of any cycle, as per investigator's discretion. After completion of treatment, participants entered follow-up phase and were not started on subsequent anti-myeloma therapy without confirmed disease progression (assessed by IMWG criteria).
Period: Overall Study
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Started | 356 | 350
Treated | 354 | 346
Completed | 0 | 0
Not Completed | 356 | 350
Not completed — Lost to Follow-up | 18 | 15
Not completed — Death | 217 | 171
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 30 | 30
Not completed — Other | 3 | 4
Not completed — Discontinued at clinical cutoff (due to end of data collection period) | 87 | 130

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP) | Total
Number analyzed (Participants) | 356 | 350 | 706
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (5.82) | 71.3 (6.66) | 71.4 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 190 | 379
  Male | 167 | 160 | 327
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 24 | 40
  Not Hispanic or Latino | 332 | 320 | 652
  Unknown or Not Reported | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 45 | 47 | 92
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 304 | 297 | 601
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 2 | 2 | 4
  Australia | 10 | 5 | 15
  Belgium | 8 | 6 | 14
  Brazil | 2 | 4 | 6
  Bulgaria | 15 | 8 | 23
  Croatia | 2 | 2 | 4
  Czech Republic | 29 | 21 | 50
  Georgia | 11 | 11 | 22
  Germany | 2 | 5 | 7
  Greece | 15 | 14 | 29
  Hungary | 12 | 14 | 26
  Italy | 26 | 28 | 54
  Japan | 26 | 24 | 50
  Poland | 27 | 39 | 66
  Portugal | 4 | 3 | 7
  Macedonia | 10 | 1 | 11
  Romania | 18 | 10 | 28
  Russia | 21 | 22 | 43
  Serbia | 3 | 7 | 10
  Korea, Republic of | 18 | 23 | 41
  Spain | 47 | 56 | 103
  Turkey | 10 | 5 | 15
  Ukraine | 20 | 28 | 48
  United Kingdom | 15 | 9 | 24
  United States | 3 | 3 | 6
Stage of Disease (ISS) [Count of Participants; unit: Participants] — The International Staging System (ISS) consists of following 3 stages - Stage I: serum beta2-microglobulin less than (<) 3.5 milligrams per liter (mg/L) and albumin greater than or equal to (>=) 3.5 grams per 100 Milliliter (g/100 mL); Stage II: neither stage I nor stage III and Stage III: serum beta2-microglobulin >= 5.5 mg/L.
  Participants
    Stage I | 67 | 69 | 136
    Stage II | 160 | 139 | 299
    Stage III | 129 | 142 | 271
Time from multiple myeloma (MM) diagnosis [Mean (Standard Deviation); unit: Months] — Time from multiple myeloma (MM) diagnosis is the time from diagnosis of multiple myeloma to randomization in each treatment group.
  Months | 1.27 (1.737) | 1.09 (1.056) | 1.18 (1.442)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS: duration from date of randomization to progressive disease (PD)/death, whichever occurs first. PD per IMWG criteria-Increase of 25% from lowest response value in one of following: Serum M-component (absolute increase >=0.5 grams per deciliter [g/dL]); Urine M-component (absolute increase >=200 milligrams [mg]/24 hours); Only participants without measurable serum and urine M-protein levels: difference between involved and uninvolved free light chain (FLC) levels (absolute increase >10 mg/dL); Only participants without measurable serum and urine M-protein levels, without measurable disease by FLC levels, bone marrow Plasma cells (PC) percentage (%) (absolute % >=10%); Bone marrow PC%: absolute% >10%; Definite development of new bone lesions/soft tissue plasmacytomas/definite increase in size of existing bone lesions/soft tissue plasmacytomas and Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the PC proliferative disorder.
Time Frame: From randomization (Day -3) up to 2.4 years
Population: Intent-to-treat (ITT) population included all participants randomized into the study; classified according to assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Months | 18.14 [16.53 to 19.91] | NA [NA to NA] — Here 'NA' signifies that median and 95% confidence interval (CI) was not estimable due to insufficient number of events.

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The Overall response rate was defined as the percentage of participants who achieved a partial response (PR) or better, according to the International Myeloma Working Group (IMWG) criteria, during the study or during follow up. IMWG criteria for PR: greater than or equal to (>=) 50 percentage (%) reduction of serum M-protein and reduction in 24 hour urinary M-protein by >=90% or to <200 mg/24 hours, if the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved free light chain (FLC) levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow plasma cells (PCs) is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%, in addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: From randomization (Day -3) up to 2.4 years
Population: ITT population included all participants randomized into the study; classified according to assigned treatment group, regardless of the actual treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Percentage of participants | 73.9 | 90.9

3. Secondary Outcome: Percentage of Participants With Very Good Partial Response (VGPR) or Better
Description: VGPR or better rate was defined as the percentage of participants who achieved VGPR or complete response (CR) (including stringent complete response[sCR]) according to the IMWG criteria during or after the study treatment. VGPR: Serum and urine component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein level less than (<) 100 milligram (mg) per 24 hour; CR: negative immunofixation on the serum and urine, Disappearance of any soft tissue plasmacytomas and < 5% plasms cells (PCs) in bone marrow; sCR: CR in addition to having a normal FLC ratio and an absence of clonal cells in bone marrow by immunohistochemistry, immunofluorescence, 2-4 color flow cytometry.
Time Frame: From randomization (Day -3) up to 2.4 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Percentage of participants | 49.7 | 71.1

4. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Better
Description: CR or better rate was defined as the percentage of participants with a CR or better (i.e. CR and sCR) as per IMWG criteria. CR: as negative immunofixation on the serum and urine and disappearance of soft tissue plasmacytomas and less than (<) 5 percent plasma cells in bone marrow; sCR: CR plus normal free light chain (FLC) ratio and absence of clonal PCs by immunohistochemistry, immunofluorescence or 2- to 4-color flow cytometry.
Time Frame: From randomization (Day -3) up to 2.4 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Percentage of participants | 24.4 | 42.6

5. Secondary Outcome: Percentage of Participants With Stringent Complete Response (sCR)
Description: sCR as per IMWG criteria is CR plus normal free light chain (FLC) ratio and absence of clonal PCs by immunohistochemistry, immunofluorescence or 2- to 4-color flow cytometry. CR: Negative immunofixation on the serum and urine; Disappearance of any soft tissue plasmacytomas; <5% plasma cells (PCs) in bone marrow.
Time Frame: From randomization (Day -3) up to 2.4 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Percentage of participants | 7.0 | 18.0

6. Secondary Outcome: Percentage of Participants With Negative Minimal Residual Disease (MRD)
Description: The Minimal Residual Disease negativity rate was defined as the percentage of participants who had negative MRD (detection of less than 1 malignant cell among 100,000 normal cells) assessment at any timepoint after the first dose of study drugs by evaluation of bone marrow aspirates or whole blood at 10^-5 threshold. MRD was evaluated by using Deoxyribonucleic acid (DNA) sequencing of immunoglobulin genes. MRD was assessed in participants who achieved complete response or stringent complete response (CR/sCR).
Time Frame: From randomization (Day -3) up to 8.3 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Percentage of participants | 7.0 [4.6 to 10.2] | 28.3 [23.6 to 33.3]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was measured from the date of randomization to date of death. Median Overall Survival was estimated by using the Kaplan-Meier method.
Time Frame: From randomization (Day -3) up to 8.3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Months | 53.59 [46.32 to 60.91] | 82.96 [72.48 to NA] — Here 'NA' signifies that upper limit of 95% CI was not estimable due to insufficient number of participants with events.

8. Secondary Outcome: Progression Free Survival on Next Line of Therapy (PFS2)
Description: Progression-free survival after next-line therapy is defined as the time from randomization to progression on the next line of subsequent antimyeloma therapy or death due to any cause (prior to start of second line of antimyeloma therapy), whichever comes first. Disease progression on next line of treatment was based on investigator judgment.
Time Frame: From randomization (Day -3) up to 8.3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Months | 42.41 [37.29 to 47.05] | 66.73 [58.58 to 80.07]

9. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP: Time from date of randomization to date of first documented evidence of PD or death due to PD, whichever occurs first. PD per IMWG criteria- Increase of 25 % from lowest response value in one of following: Serum M-component (absolute increase >=0.5 g/dL); Urine M-component (absolute increase >=200 mg/24 hours); Only in participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase >10 milligram per deciliter [mg/dL]); Only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow plasma cells (PC)% (absolute % >=10%); Bone marrow PC %: absolute % >10%; Definite development of new bone lesions/soft tissue plasmacytomas or definite increase in size of existing bone lesions/soft tissue plasmacytomas and Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the PC proliferative disorder.
Time Frame: From randomization (Day -3) up to 2.4 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Months | 19.35 [17.38 to 22.67] | NA [NA to NA] — Here 'NA' signifies that median and 95% CI was not estimable due to insufficient number of events.

10. Secondary Outcome: Time to Response
Description: Time to response, defined as the time between the date of randomization and the first efficacy evaluation that the participant has met all criteria for PR or better. PR: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours; If the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria; If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow PCs is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: From randomization (Day -3) up to 2.4 years
Population: Response-evaluable population: participants who have a confirmed diagnosis of MM and measurable disease at baseline or screening, must receive at least one component of study treatment and have adequate post-baseline disease assessments. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this endpoint.
Measure: Median (Full Range); unit: Months
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 263 | 318
Months | 0.82 [0.7 to 12.6] | 0.79 [0.4 to 15.5]

11. Secondary Outcome: Duration of Response (DOR)
Description: DOR: participants with confirmed response (PR or better) as time between first documentation of response and disease progression per IMWG response criteria, or death due to PD, whichever occurs first. PD: Increase of 25% from lowest response value in any one of following: Serum M-component (absolute increase>=0.5 g/dL); Urine M-component (absolute increase>=200 mg/24 hours); Only participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase >10mg/dL); Only participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC%(absolute%>=10%); Bone marrow PC's %: absolute%>10%; Definite development of new bone lesions/soft tissue plasmacytomas/definite increase in the size of existing bone lesions or soft tissue plasmacytomas and Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: From first documentation of response up to 2.4 years
Population: Response-evaluable set: participants who have a confirmed diagnosis of MM and measurable disease at baseline or screening. Participants must have received at least one component of study treatment and have adequate post-baseline disease assessments. Here 'N'(overall number of participants analyzed) signifies number of participants evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 263 | 318
Months | 21.3 [18.4 to NA] — Here 'NA' signifies that upper limit of 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here 'NA' signifies that median and 95% CI was not estimable due to insufficient number of events.

12. Secondary Outcome: Time to Next Treatment (TNT)
Description: Time to next treatment is defined as the time from randomization to the start of the next-line treatment. Kaplan-Meier method was used for the analysis.
Time Frame: From randomization (Day -3) up to 8.3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Months | 25.9 [23.4 to 28.6] | 66.8 [47.9 to NA] — Here 'NA' signifies that upper limit of 95% CI was not estimable due to insufficient number of events.

13. Secondary Outcome: Percentage of Participants With Best M-protein Response
Description: Percentage of participants with Best M- protein response of 100% reduction and >=90% to < 100% reduction were assessed. Best M-protein response was defined as the maximal percent reduction or the lowest percent increase from baseline in serum M-protein for participants with measurable heavy chain at baseline or urine M-protein for participants without measurable heavy chain, but with measurable light chain disease at baseline. For participants without measurable heavy chain and light chain disease at baseline, best response in serum free light chain (FLC) was defined as the maximal percent reduction or the lowest percent increase from baseline in the difference between involved and uninvolved serum FLC level (dFLC).
Time Frame: Up to 2.4 years
Population: Response-evaluable set: participants have confirmed diagnosis of MM and measurable disease at baseline or screening. Participants must receive at least one component of study treatment, have adequate post-baseline disease assessments. Here, 'n' (number analyzed) signifies number of participants analyzed for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 341 | 337
Percentage of participants
  Best M-protein response in serum: 100% reduction: number analyzed (Participants) | 287 | 277
  Best M-protein response in serum: 100% reduction | 38.7 | 58.5
  Best M-protein response in serum:>= 90 to < 100%: number analyzed (Participants) | 287 | 277
  Best M-protein response in serum:>= 90 to < 100% | 14.6 | 15.2
  Best M-protein response in urine:100% reduction: number analyzed (Participants) | 36 | 42
  Best M-protein response in urine:100% reduction | 69.4 | 90.5
  Best M-protein response in urine:>=90 to < 100%: number analyzed (Participants) | 36 | 42
  Best M-protein response in urine:>=90 to < 100% | 13.9 | 7.1
  Best response in dFLC:100% reduction: number analyzed (Participants) | 18 | 18
  Best response in dFLC:100% reduction | 0 | 0
  Best response in dFLC: >=90% to < 100% reduction: number analyzed (Participants) | 18 | 18
  Best response in dFLC: >=90% to < 100% reduction | 77.8 | 100.0

14. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30: Emotional Functioning Score
Description: The EORTC QLQ-C30 is a 30 items self-reporting questionnaire, with a 1 week recall period, resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 Global Health Status (GHS) scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The questionnaire includes 28 items with 4-point Likert type responses from "1-not at all" to "4-very much" to assess functioning and symptoms; 2 items with 7-point Likert scales (1= poor and 7= excellent) for global health and overall QoL. Scores are transformed to a 0 to 100 scale, with higher scores representing better GHS, better functioning, and more symptoms. Negative change from baseline values for function and GHS scale indicated deterioration in quality of life or functioning and positive values indicate improvement.
Time Frame: Baseline (Day -24), Months 3, 6, 9, 12 ,18, 24, 30, 36, 42 and 48
Population: ITT population: participants randomized into the study; classified according to assigned treatment group, regardless actual treatment received. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants who were analyzed at each specified timepoint, for each arm, respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 327 | 317
Units on a scale
  Month 3: number analyzed (Participants) | 245 | 262
  Month 3 | 9.4 [7.1 to 11.6] | 8.5 [6.3 to 10.7]
  Month 6: number analyzed (Participants) | 213 | 235
  Month 6 | 10.5 [8.1 to 12.9] | 10.8 [8.6 to 13.1]
  Month 9: number analyzed (Participants) | 189 | 228
  Month 9 | 11.8 [9.4 to 14.3] | 11.1 [8.8 to 13.4]
  Month 12: number analyzed (Participants) | 185 | 222
  Month 12 | 11.2 [8.7 to 13.7] | 12.6 [10.3 to 14.9]
  Month 18: number analyzed (Participants) | 136 | 195
  Month 18 | 12.8 [10.1 to 15.6] | 12.5 [10.1 to 14.9]
  Month 24: number analyzed (Participants) | 83 | 152
  Month 24 | 11.8 [8.5 to 15.1] | 10.7 [8.2 to 13.3]
  Month 30: number analyzed (Participants) | 71 | 159
  Month 30 | 10.8 [7.3 to 14.3] | 12.4 [9.8 to 14.9]
  Month 36: number analyzed (Participants) | 48 | 145
  Month 36 | 10.8 [6.7 to 14.9] | 12.3 [9.6 to 14.9]
  Month 42: number analyzed (Participants) | 33 | 125
  Month 42 | 6.5 [1.7 to 11.4] | 12.8 [10 to 15.6]
  Month 48: number analyzed (Participants) | 23 | 102
  Month 48 | 6.2 [0.5 to 11.9] | 10.5 [7.5 to 13.5]

15. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30: Global Health Scale
Description: as for outcome 14
Time Frame: Baseline (Day -24), Months 3, 6, 9, 12 ,18, 24, 30, 36, 42 and 48
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 327 | 317
Units on a scale
  Month 3: number analyzed (Participants) | 245 | 262
  Month 3 | 4 [1.7 to 6.3] | 7.5 [5.2 to 9.7]
  Month 6: number analyzed (Participants) | 213 | 235
  Month 6 | 8.8 [6.4 to 11.3] | 8.5 [6.2 to 10.8]
  Month 9: number analyzed (Participants) | 189 | 228
  Month 9 | 10.2 [7.7 to 12.8] | 10.6 [8.2 to 12.9]
  Month 12: number analyzed (Participants) | 185 | 222
  Month 12 | 10.7 [8.2 to 13.3] | 11.4 [9 to 13.7]
  Month 18: number analyzed (Participants) | 136 | 195
  Month 18 | 11.8 [9 to 14.6] | 12.8 [10.3 to 15.3]
  Month 24: number analyzed (Participants) | 83 | 152
  Month 24 | 11.5 [8.1 to 15] | 9.5 [6.8 to 12.1]
  Month 30: number analyzed (Participants) | 71 | 159
  Month 30 | 10.8 [7.1 to 14.5] | 11.8 [9.2 to 14.5]
  Month 36: number analyzed (Participants) | 48 | 145
  Month 36 | 8.6 [4.2 to 12.9] | 11.9 [9.1 to 14.6]
  Month 42: number analyzed (Participants) | 33 | 125
  Month 42 | 4.8 [-0.3 to 9.9] | 10.4 [7.5 to 13.3]
  Month 48: number analyzed (Participants) | 23 | 102
  Month 48 | 8.9 [2.8 to 14.9] | 9.8 [6.6 to 12.9]

16. Secondary Outcome: Change From Baseline in EuroQol-5 Dimensions-5 Levels (EQ-5D-5L): Visual Analogue Scale (VAS)
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L Visual Analog Scale. The Visual Analogue Scale is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Baseline (Day- 24), Months 3, 6, 9, 12 ,18, 24, 30, 36, 42 and 48
Population: ITT population: participants randomized into the study; classified according to assigned treatment group, regardless actual treatment received. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants who were analyzed at each specified timepoint, for each arm, respectively. n=0 indicated that no participant was available for assessment at specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 325 | 315
Units on a scale
  Month 3: number analyzed (Participants) | 242 | 258
  Month 3 | 4.27 (18.38) | 9.37 (20.222)
  Month 6: number analyzed (Participants) | 210 | 230
  Month 6 | 7.51 (17.957) | 11.02 (20.168)
  Month 9: number analyzed (Participants) | 185 | 227
  Month 9 | 10.08 (19.475) | 12.51 (20.564)
  Month 12: number analyzed (Participants) | 185 | 217
  Month 12 | 11.1 (19.139) | 10.93 (20.447)
  Month 18: number analyzed (Participants) | 134 | 194
  Month 18 | 10.75 (21.146) | 15.35 (21.168)
  Month 24: number analyzed (Participants) | 82 | 150
  Month 24 | 10.62 (19.531) | 12.17 (22.592)
  Month 30: number analyzed (Participants) | 71 | 157
  Month 30 | 12.38 (21.817) | 14.41 (21.305)
  Month 36: number analyzed (Participants) | 46 | 143
  Month 36 | 12 (23.856) | 13.94 (21.984)
  Month 42: number analyzed (Participants) | 33 | 123
  Month 42 | 12.88 (23.789) | 14.33 (21.502)
  Month 48: number analyzed (Participants) | 23 | 99
  Month 48 | 9.17 (18.612) | 11.93 (24.031)

17. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions-5 Level (EQ-5D-5L) Utility Score
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L Visual Analog Scale. The EQ-5D-5L descriptive system provides a profile of the participant's health state 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The participant was asked to indicate his/her current health state by selecting the most appropriate level in each of the 5 dimensions. Responses to the 5 dimension scores were combined and converted into a single preference-weighted health utility index score 0 (0.0- worst health state) to 1 (1.0- better health state) representing the general health status of the individual based on the UK scoring algorithm.
Time Frame: Baseline (Day -24), Months 3, 6, 9, 12 ,18, 24, 30, 36, 42 and 48
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 325 | 315
Units on a scale
  Month 3: number analyzed (Participants) | 242 | 258
  Month 3 | 0.09 (0.312) | 0.12 (0.266)
  Month 6: number analyzed (Participants) | 210 | 230
  Month 6 | 0.12 (0.269) | 0.14 (0.271)
  Month 9: number analyzed (Participants) | 185 | 227
  Month 9 | 0.16 (0.27) | 0.16 (0.271)
  Month 12: number analyzed (Participants) | 185 | 217
  Month 12 | 0.15 (0.281) | 0.17 (0.288)
  Month 18: number analyzed (Participants) | 134 | 194
  Month 18 | 0.14 (0.268) | 0.17 (0.293)
  Month 24: number analyzed (Participants) | 82 | 150
  Month 24 | 0.15 (0.252) | 0.18 (0.312)
  Month 30: number analyzed (Participants) | 71 | 157
  Month 30 | 0.16 (0.291) | 0.19 (0.303)
  Month 36: number analyzed (Participants) | 47 | 143
  Month 36 | 0.16 (0.315) | 0.21 (0.306)
  Month 42: number analyzed (Participants) | 33 | 123
  Month 42 | 0.08 (0.303) | 0.2 (0.287)
  Month 48: number analyzed (Participants) | 23 | 99
  Month 48 | 0.07 (0.246) | 0.15 (0.319)

18. Post Hoc Outcome: Progression Free Survival at Data Cutoff Date of 24 June 2019
Description: PFS: duration from date of randomization to PD/death, whichever occurs first. PD per IMWG criteria-Increase of 25% from lowest response value in one of following: Serum M-component (absolute increase >=0.5 g/dL); Urine M-component (absolute increase >=200 mg/24 hours); Only participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase >10 mg/dL); Only participants without measurable serum and urine M-protein levels, without measurable disease by FLC levels, bone marrow PC %(absolute % >=10%); Bone marrow PC %: absolute % >10 %; Definite development of new bone lesions/soft tissue plasmacytomas/definite increase in size of existing bone lesions/soft tissue plasmacytomas and development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the PC proliferative disorder.
Time Frame: From randomization (Day -3) up to 4.4 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
Number analyzed (Participants) | 356 | 350
Months | 19.29 [17.97 to 20.40] | 36.40 [32.13 to 45.90]

ADVERSE EVENTS:
Time Frame: All cause mortality: From randomization (Day -3) up to 8.3 years; Serious and Other AEs: From start of treatment (Day 1) up to 30 days after last dose of study treatment (up to 8.2 years)
Description: All cause mortality: All participants randomized into the study. Serious and Other AEs: Safety population defined as participants who had received at least 1 administration of any study treatment (partial or complete) and were analyzed according to treatment actually received.
Arm/Group | Velcade, Melphalan and Prednisone (VMP) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP)
All-Cause Mortality (participants affected / at risk) | 217/356 | 172/350
Serious Adverse Events (participants affected / at risk) | 117/354 | 186/346
Other Adverse Events (participants affected / at risk) | 331/354 | 329/346
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade, Melphalan and Prednisone (VMP) (N=354) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP) (N=346)
Anaemia (Blood and lymphatic system disorders) | 9 | 8
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 6
Acute Coronary Syndrome (Cardiac disorders) | 1 | 2
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 5
Angina Pectoris (Cardiac disorders) | 0 | 2
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 6
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 2 | 1
Cardiac Failure (Cardiac disorders) | 8 | 2
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Cardiac Failure Chronic (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 2
Myocardial Infarction (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 2
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1
Stress Cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Hypertrophic Cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Conjunctival Haemorrhage (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 1
Abdominal Adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 | 1
Acute Abdomen (Gastrointestinal disorders) | 0 | 1
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Appendiceal Mucocoele (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Diverticular Perforation (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 2
Femoral Hernia (Gastrointestinal disorders) | 0 | 1
Gastric Dilatation (Gastrointestinal disorders) | 0 | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal Rupture (Gastrointestinal disorders) | 1 | 0
Oesophagitis Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Rectal Polyp (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 2
Asthenia (General disorders) | 2 | 2
Chest Pain (General disorders) | 0 | 1
Death (General disorders) | 2 | 2
Fatigue (General disorders) | 2 | 1
Generalised Oedema (General disorders) | 0 | 2
Hyperthermia (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 5 | 5
Strangulated Hernia (General disorders) | 0 | 1
Sudden Death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 10
Candida Sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Colitis (Infections and infestations) | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 2 | 0
Covid-19 (Infections and infestations) | 0 | 5
Covid-19 Pneumonia (Infections and infestations) | 0 | 3
Cytomegalovirus Infection (Infections and infestations) | 0 | 1
Cytomegalovirus Infection Reactivation (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Enterococcal Bacteraemia (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 1
Escherichia Bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
H1n1 Influenza (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Herpes Zoster Disseminated (Infections and infestations) | 0 | 1
Infected Fistula (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 3
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 0
Infective Myositis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 5
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 10
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Meningitis Pneumococcal (Infections and infestations) | 0 | 1
Neutropenic Infection (Infections and infestations) | 1 | 1
Pelvic Infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Pneumococcal Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 13 | 53
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Pneumonia Pneumococcal (Infections and infestations) | 0 | 3
Pneumonia Streptococcal (Infections and infestations) | 1 | 0
Pneumonia Viral (Infections and infestations) | 0 | 2
Postoperative Abscess (Infections and infestations) | 0 | 1
Pseudomembranous Colitis (Infections and infestations) | 0 | 1
Pulmonary Sepsis (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 5 | 6
Septic Shock (Infections and infestations) | 2 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Tuberculous Pleurisy (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 7
Urinary Tract Infection (Infections and infestations) | 1 | 5
Urinary Tract Infection Bacterial (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Varicella Zoster Virus Infection (Infections and infestations) | 0 | 1
Vascular Device Infection (Infections and infestations) | 1 | 1
Wound Infection (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Chest Injury (Injury, poisoning and procedural complications) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 2
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 4
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Heart Injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 2 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic Bone Injury (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 5
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 2
Traumatic Shock (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 2
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 0
Blood Creatinine Increased (Investigations) | 1 | 1
C-Reactive Protein Increased (Investigations) | 0 | 2
Oxygen Saturation Decreased (Investigations) | 0 | 2
Troponin Increased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Autonomic Nervous System Imbalance (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Ischaemic Stroke (Nervous system disorders) | 1 | 3
Neuralgia (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Parkinson's Disease (Nervous system disorders) | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 2
Sciatica (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Agitation (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 5 | 3
Anuria (Renal and urinary disorders) | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Prerenal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 2
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Hypertensive Crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Hypovolaemic Shock (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade, Melphalan and Prednisone (VMP) (N=354) | Daratumumab, Velcade, Melphalan and Prednisone (D-VMP) (N=346)
Anaemia (Blood and lymphatic system disorders) | 129 | 110
Leukopenia (Blood and lymphatic system disorders) | 53 | 47
Lymphopenia (Blood and lymphatic system disorders) | 36 | 39
Neutropenia (Blood and lymphatic system disorders) | 186 | 174
Thrombocytopenia (Blood and lymphatic system disorders) | 189 | 172
Atrial Fibrillation (Cardiac disorders) | 7 | 20
Abdominal Pain (Gastrointestinal disorders) | 25 | 26
Abdominal Pain Upper (Gastrointestinal disorders) | 13 | 21
Constipation (Gastrointestinal disorders) | 64 | 64
Diarrhoea (Gastrointestinal disorders) | 87 | 100
Dyspepsia (Gastrointestinal disorders) | 12 | 22
Nausea (Gastrointestinal disorders) | 76 | 76
Vomiting (Gastrointestinal disorders) | 52 | 62
Asthenia (General disorders) | 43 | 51
Chills (General disorders) | 6 | 28
Fatigue (General disorders) | 50 | 60
Influenza Like Illness (General disorders) | 5 | 18
Injection Site Erythema (General disorders) | 28 | 12
Oedema Peripheral (General disorders) | 39 | 68
Pyrexia (General disorders) | 70 | 87
Bronchitis (Infections and infestations) | 25 | 71
Covid-19 (Infections and infestations) | 0 | 25
Herpes Zoster (Infections and infestations) | 12 | 22
Influenza (Infections and infestations) | 10 | 23
Nasopharyngitis (Infections and infestations) | 22 | 50
Pneumonia (Infections and infestations) | 7 | 39
Respiratory Tract Infection (Infections and infestations) | 1 | 22
Upper Respiratory Tract Infection (Infections and infestations) | 48 | 103
Urinary Tract Infection (Infections and infestations) | 13 | 43
Alanine Aminotransferase Increased (Investigations) | 17 | 23
Aspartate Aminotransferase Increased (Investigations) | 13 | 19
Decreased Appetite (Metabolism and nutrition disorders) | 46 | 42
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 26
Hypocalcaemia (Metabolism and nutrition disorders) | 18 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 49
Back Pain (Musculoskeletal and connective tissue disorders) | 40 | 67
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 27
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 11 | 18
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 10 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 18
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 22 | 40
Dizziness (Nervous system disorders) | 21 | 33
Headache (Nervous system disorders) | 12 | 35
Neuralgia (Nervous system disorders) | 16 | 26
Paraesthesia (Nervous system disorders) | 19 | 23
Peripheral Sensory Neuropathy (Nervous system disorders) | 122 | 100
Insomnia (Psychiatric disorders) | 32 | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 70
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 43
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 28
Rash (Skin and subcutaneous tissue disorders) | 49 | 40
Hypertension (Vascular disorders) | 10 | 50
Hypotension (Vascular disorders) | 23 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT02195479/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT02195479/SAP_001.pdf